CLINICAL TRIAL: NCT01475760
Title: A Multi-Center, Open Label Study to Evaluate Chitosan Chewing Gum in Patients With Chronic Kidney Disease
Brief Title: A Study to Evaluate Chitosan Chewing Gum in Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Nephrologists, P.C. (Other)
Collaborators: CM&D Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CMD007
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; serum phosphorus; salivary phosphorus; FGF23
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Chitosan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- K2CG chewing gum (20 mg chitosan) (Active Comparator)
  Interventions: Other: K2CG chewing gum (20mg chitosan)
- K2CG chewing gum (60 mg chitosan) (Active Comparator)
  Interventions: Other: K2CG chewing gum (60mg chitosan)
- Standard of Care (No Intervention)

INTERVENTIONS:
Other: K2CG chewing gum (20mg chitosan) — All participating subjects will chew gum TID for 14 days beginning on Day 1 through Day 14
  Arms: K2CG chewing gum (20 mg chitosan)
Other: K2CG chewing gum (60mg chitosan) — Subjects will be randomized in a 1:1 fashion to either chew gum or continue with Standard of Care (no intervention)if they have a change in serum phosphorus of greater than or equal to -0.2 mg/dL from:
  Baseline (defined as the mean of values from Visit 2, 3, and 4) to the end of active treatment (defined as the mean of Visit 6 and 7) AND/OR Baseline (defined as the mean of values from Visit 2, 3, and 4) and end of wash out (defined as Visit 7 (Day 22).
  If randomized: Chew gum TID for 14 days beginning on Day 29 through Day 42
  Arms: K2CG chewing gum (60 mg chitosan)

SUMMARY:
The purpose of this study is to determine the efficacy of chitosan chewing gum (K2CG) in reducing serum phosphorus in subjects with chronic kidney disease.

DETAILED DESCRIPTION:
Given the public health importance of increased P levels in the general population and specifically in patients with chronic kidney disease, it is of great importance to evaluate the ability of a medical food such as K2CG to reduce elevated serum P levels. In patients with CKD receiving dialysis it has been estimated that sustained control of serum P may result in an approximate 17% reduction in mortality.

The investigators have conducted a previous pilot double blind randomized controlled study of K2CG 20 mg and 40 mg BID for 4 weeks in 90 patients with ESRD. In this initial study the investigators did not observe a statistically significant reduction in either serum P or salivary P with active therapy as compared to placebo. However, a clear trend towards a reduction in serum P was seen in the randomized phase of the study with the active gum administered twice a day. During the open-label period where the gum was administered thrice-daily the investigators did see a statistically significant reduction in serum P of 0.3 mg/dL. Moreover, in patients with CKD not on dialysis, the investigators observed a reduction in mean serum P of approximately 0.2 mg/dL. While not statistically significant, this trial was not powered to detect this level of change in serum P and was underpowered to do so.. Differences in this range (0.2-0.4 mg/dL) have been reported in studies utilizing dietary manipulation (plant protein versus animal protein) and with the use of Niacin and are felt to be clinically meaningful reductions.

The investigators have previously also conducted a cross-sectional observational study evaluating salivary P levels across a wide spectrum of eGFR. The data indicate that mean salivary P is uniformly increased (15-25 mg/dL) relative to serum P (2.5- 4.5 mg/dL) being approximately 5-7X higher as shown below (group 1 = eGFR > 90, group 7= eGFR < 15). Importantly, salivary P was similar across the entire spectrum of eGFR.

The investigators have previously conducted a clinical trial evaluating several different formulations of K2CG with varying amounts of chitosan loading into the gum base, variable weights of gum base and 2 different formulations of gum base. In these trials the investigators further studied the effects of gum chewing in either the fasted or fed state and the effects of varying amounts of gum chewing time. Results from this study have demonstrated that the maximal amount of P loading into the K2CG is seen with the 1g chewing gum containing 20 mg chitosan and that the maximal effect is seen with 30 minutes of gum chewing.

Based on data from this study the investigators have chosen this strength/formulation for the primary efficacy endpoint assessment in the current protocol. Similar efficacy results with regard to total P loading per chewing gum were seen with the 2.0 gram, 60 mg chitosan chewing gum and there was an indication that subjects had a subjective preference for this formulation. As a result, this protocol will also assess (as a secondary efficacy endpoint) the reduction in serum P with this strength/formulation during an open label phase only in those subjects who have responded during the primary efficacy assessment phase. This will allow a comparison of efficacy between the 2 gum sizes/strengths among known 'responders' with regard to serum P reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women > 18 years of age;
2. The subject has voluntarily signed and dated the most recent informed consent form approved by an Institutional Review Board (IRB);
3. The subject will, in the opinion of the investigator, be compliant with prescribed therapy and all study visits;
4. Subject must be able to communicate and be able to understand and comply with the requirements of the study;
5. For subjects not on dialysis estimated GFR at screening < or equal to 60 ml/min + 10 % that in the opinion of the investigator is stable and not expected to initiate dialysis within 3 months;
6. Subject must have serum phosphorus at screening of greater than or equal to 3.5 mg/dL;
7. Subjects must have a screening salivary flow rate by Saxon test ≥ 1 g/2 min;
8. All subjects must have NO change in prescribed dose or frequency of any of the following medications ≥ 14 days prior to Run-In Visit 2 (Day -15):

a. Phosphate binding products including prescribed and over-the counter b. Oral or injectable active vitamin D c. Oral nutritional vitamin D d. Calcium supplements e. Anti-osteoporotic medication (e.g. bisphosphonates) f. Cinacalcet i. Subject must be prescribed a diet appropriate for patients with their stage of CKD, must be willing to avoid intentional changes in diet and must have stable nutritional status in the opinion of the investigator.

j. Subjects on dialysis must, in the opinion of the investigator, have a stable dialysis prescription, stable dialysis access and a URR >/= 65% for at least 4 weeks prior to Day -15.

Exclusion Criteria:

1. Subject is receiving or has received an investigational product (or is currently using an investigational device) within 14 days prior to Visit 2 (Day -15);
2. Subject has a known sensitivity to chitin or allergy to shellfish;
3. Subject has had dental work other than cleaning, cavity filling or crown placement within 48 hours prior to Visit 4 (Day 1) or at any time during the course of the trial;
4. Subject has a clinically significant infection requiring treatment with antibiotics (within 7 days prior to Visit 2 (Day -15));
5. Subject has had an inpatient hospitalization within 14 days prior to Visit 2 (Day -15) with the exception of hospitalizations related to vascular access procedures;
6. Subject has a known history of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result;
7. Active drug or alcohol dependence or abuse (excluding tobacco use) in the opinion of the principal investigator;
8. In the opinion of the investigator, subject is unable to chew gum for 30 minutes;
9. Subject has an unstable medical condition which in the opinion of the investigator would compromise successful completion of the study;
10. Subject is receiving calcimimetic therapy (acceptable if subject is on dialysis);
11. Subject has known salivary gland dysfunction or Sjogren's syndrome;
12. Subjects is receiving niacin therapy within 7 days prior to Run- In Visit 2(Day -15) (use as part of standard multivitamin is acceptable);
13. Subject has had a major cardiovascular event within 90 days of screening. The investigator should be guided by evidence of any of the following;

a. Acute myocardial infarction b. Acute cerebral vascular event c. Vascular surgical intervention d. Coronary Revascularization e. Decompensated congestive heart failure

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
serum phosphorus | change from baseline to mean during 2 weeks active therapy
  Change in serum phosphorus from baseline to mean of values during 2 week active chewing period in patients with CKD not on dialysis

SECONDARY OUTCOMES:
serum phosphorus | change from baseline after 2 weeks active chewing
  change in serum phosphorus from baseline to mean of values during active therapy in patients with CKD on dialysis
salivary phosphorus | change from baseline to mean during active therapy -2 weeks
  change in salivary phosphorus from baseline to mean of values during 2 weeks active

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Block, MD, Principal Investigator — DenverNephrologists, P.C.
Locations (4):
- United States (4):
  - Southwest Clinical Reserach Institute, LLC, Tempe, Arizona
  - Denver Nephrologists, PC, Denver, Colorado
  - Pacific Renal Research Institute, Meridian, Idaho
  - Renal Associates, PA, San Antonio, Texas

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Block GA, Persky MS, Shamblin BM, Baltazar MF, Singh B, Sharma A, Pergola P, Smits G, Comelli MC. Effect of salivary phosphate-binding chewing gum on serum phosphate in chronic kidney disease. Nephron Clin Pract. 2013;123(1-2):93-101. doi: 10.1159/000351850. Epub 2013 Jun 22. PMID 23797006